CLINICAL TRIAL: NCT00684190
Title: An Open, Randomised, Three Period Cross, Single Centre, Phase 1 Pharmacokinetic Interaction Study of the Reflux Inhibitor AZD3355 150 mg Bid and Esomeprazole 40 mg od After 7 Days of Treatment in Healthy Volunteers
Brief Title: Drug Interaction Study Between AZD3355 and Nexium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Debra G. Silberg, MD, PhD, Medical Science Director, AZD3355, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D9120C00016; EudraCt nr 2007-007128-16
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Reflux Inhibitor; GERD; PPI Interaction
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AZD3355 150 mg
  Interventions: Drug: AZD3355
- 2 (Experimental): Esomeprazole 40mg
  Interventions: Drug: Esomeprazole
- 3 (Experimental): AZD3355 150mg/Esomeprazole 40mg
  Interventions: Drug: AZD3355; Drug: Esomeprazole

INTERVENTIONS:
Drug: AZD3355 — 150 mg bid, oral, 7 days
  Other Names: Lesogaberan
  Arms: 1; 3
Drug: Esomeprazole — 40 mg od, oral, 7 days
  Other Names: Nexium
  Arms: 2; 3

SUMMARY:
The purpose of the study is to evaluate if AZD3355 and Nexium interact with each other or not, i.e. show the same or altered plasma concentration profiles when co-administered compared to administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Females no childbearing potential
* Clinically normal physical findings

Exclusion Criteria:

* Clinically significant illness within 2 weeks prior to the first dose of investigational product
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during day 7 each treatment period

SECONDARY OUTCOMES:
4-BOH cholesterol | Sampling occasions during day 7 one treatment period (AZD3355 alone)
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ersdal, PhD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Jan Vouis, MD, Principal Investigator — Quintiles AB, Uppsala, Sweden
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Derived] Niazi M, Silberg DG, Miller F, Ruth M, Holmberg AA. Evaluation of the pharmacokinetic interaction between lesogaberan (AZD3355) and esomeprazole in healthy subjects. Drugs R D. 2010;10(4):243-51. doi: 10.2165/11588180-000000000-00000. PMID 21171670